CLINICAL TRIAL: NCT00466297
Title: The SCRIPT Programme (GIM): Structuring Communication Relationships for Interprofessional Teamwork to Achieve Interprofessional Education for Collaborative Patient-Centered Practice (IECPCP)
Brief Title: Interprofessional Collaborative Communication in Acute Care Hospital Teams
Acronym: SCRIPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Health Canada (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Health Canada 102117
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2007-04

CONDITIONS: Disease; Delivery of Healthcare
Keywords: Interprofessional; Collaboration; Teamwork; General internal medicine; Cluster randomized
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Face-to-face communication interactions

SUMMARY:
Collaborative practice may improve patient outcomes in specific disease conditions and health care settings. The SCRIPT Programme is an intervention to implement informal, but structured, communication etiquette between members of interprofessional ward-based clinical teaching units (CTUs) in General Internal Medicine (GIM) hospital divisions.

DETAILED DESCRIPTION:
A recent literature review commissioned by Health Canada for the Inter-Professional Education for Collaborative Patient-Centred Practice initiative (IECPCP) reported evidence that collaborative practice improves patient outcomes in specific populations. Interprofessional collaborative teaching and practicing are poorly articulated in the literature, however. Studies are needed that can develop a trial-based body of evidence to support education and practice of effective interprofessional care.

The SCRIPT project will attempt to develop sustainable transformation in the conduct, learning and evaluation of interprofessional teamwork in the Toronto Academic Health Science Network (TAHSN). SCRIPT has investigated interprofessional work relations in general internal medicine units at TAHSN hospitals using fieldwork observations and interview methods. These data were foundational for SCRIPT's design of a unit-based staff intervention intended to promote more--and more-effective--informal interprofessional communication and collaboration between GIM staff members outside of traditional, structured meeting times like morning report and bullet rounds.

The intervention is designed as part of a pragmatic trial. We will ask GIM division staff of intervention teams to implement a 4-step communication protocol in face-to-face, patient-related interaction. The steps are:

1. introduce oneself by name;
2. state one's role or responsibility in relation to the patient under discussion;
3. describe the issue, problem, or plan relating to the target patient;
4. elicit feedback from the other participant(s) in the interaction with a prompt, e.g., "do you have any concerns," or, "is there something else I should consider?"

The intervention will be evaluated as a cluster randomized controlled trial among five large Toronto (Canada) teaching hospitals. Two medical clinical teaching units and associated ward teams of nurses and other health professionals from each hospital's GIM division will be allocated at random to enact the intervention. Two other GIM CTUs in each hospital will continue their usual interprofessional practice, without intervention. In total, there are 20 CTUs, 10 in the treatment group and 10 in the control group. Intervention CTUs will be compared with control CTUs on the outcomes of interest.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to divisions of General Internal Medicine
* Health care providers working in divisions of General Internal Medicine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2007-04; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
unplanned hospital readmission 7 days post-discharge and 30 days post-discharge

SECONDARY OUTCOMES:
length of stay in hospital for GIM patients' index admission
measurement survey of staff members' perceptions of interprofessional collaboration
patient satisfaction measured by a large standardized, cross-site survey regime
calls placed to staff members' paging devices
use of evidence-based, optimal prescription drug therapy

CONTACTS AND LOCATIONS:
Overall Officials: Merrick Zwarenstein, MB BCh, MS, Principal Investigator — Institute for Clinical Evaluative Sciences, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

REFERENCES:
- [Background] Reeves S, Russell A, Zwarenstein M, Kenaszchuk C, Conn LG, Doran D, Sinclair L, Lingard L, Oandasan I, Thorpe K, Austin Z, Beales J, Hindmarsh W, Whiteside C, Hodges B, Nasmith L, Silver I, Miller KL, Vogwill V, Strauss S. Structuring communication relationships for interprofessional teamwork (SCRIPT): a Canadian initiative aimed at improving patient-centred care. J Interprof Care. 2007 Feb;21(1):111-4. doi: 10.1080/13561820600991595. No abstract available. PMID 17365378
- [Derived] Zwarenstein M, Reeves S, Russell A, Kenaszchuk C, Conn LG, Miller KL, Lingard L, Thorpe KE. Structuring Communication Relationships for Interprofessional Teamwork (SCRIPT): a cluster randomized controlled trial. Trials. 2007 Sep 18;8:23. doi: 10.1186/1745-6215-8-23. PMID 17877830